CLINICAL TRIAL: NCT02086370
Title: Prophylactic Salpingectomy for the Prevention of the Ovarian Cancer: Comparison Between Surgical Techniques. A Randomized Controlled Trial
Brief Title: Prophylactic Salpingectomy for the Prevention of the Ovarian Cancer: Comparison Between Surgical Techniques
Acronym: Rad_PBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Fulvio Zullo, Full Professor Obstetric Gynecology, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Radical_PBS
Record Dates: First submitted 2014-03-09; First posted 2014-03-13 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Uterine Fibroids; Contraception Desired
Keywords: PBS; Prophylactic bilateral salpingectomy; Ovarian cancer prevention; Ovarian reserve; Permanent contraception; Surgical sterilization
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard PBS (Active Comparator): the tube will be removed by coagulation and section of the tissue beginning from the very distal fimbrial and proceeding toward the uterine cornu. The resection will be performed at the level of the posterior tubal margin, sparing the mesosalpinx
  Interventions: Procedure: Standard PBS
- Radical PBS (Experimental): the tube will be removed by coagulation and section of the tissue beginning from the very distal fimbrial and proceeding toward the uterine cornu. The resection will be performed at the level of ovarian margin and the uterus-ovarian ligament, including the mesosalpinx removal
  Interventions: Procedure: Radical PBS

INTERVENTIONS:
Procedure: Standard PBS — the tube will be removed by coagulation and section of the tissue beginning from the very distal fimbrial and proceeding toward the uterine cornu. The resection will be performed at the level of the posterior tubal margin, sparing the mesosalpinx.
  Arms: Standard PBS
Procedure: Radical PBS — the tube will be removed by coagulation and section of the tissue beginning from the very distal fimbrial and proceeding toward the uterine cornu. The resection will be performed at the level of ovarian margin and the uterus-ovarian ligament, including the mesosalpinx removal.
  Arms: Radical PBS

SUMMARY:
The aim of this RCT of study is to compare the outcomes of the standard salpingectomy (removal of the fallopian tube) with the radical removal of the tube and the mesosalpinx in terms of ovarian reserve.

DETAILED DESCRIPTION:
Ovarian cancer accounts for 3% of all female cancers and represents the fifth leading cause of cancer death in the Western world (1). In 90% of cases, these are epithelial ovarian cancers (2).

Because of the biological aggressiveness of this tumor and nonspecific symptoms, that causes a diagnosis at an advanced stage in 75% of cases, ovarian cancer is the gynecological cancer with the highest mortality rate (3).

To date, an effective screening strategy to the early diagnosis of ovarian cancer doesn't exist, so the prophylactic adnexectomy is the only available tool to reduce the incidence and the mortality rate, even if the role of this surgical strategy is controversial, especially in premenopausal women (4). In fact, the American College of Obstetricians and Gynaecologists (ACOG) guidelines recommend the ovarian preservation in premenopausal women with no family history or other risk factors for ovarian cancer (5).

Some clinical studies have shown that the prophylactic adnexectomy and the consequent surgical menopause increase significantly the long term risk of cardiovascular and psychosexual diseases. (6-8). In particular, a case-control study done in a population of 29,380 women subjected to hysterectomy with and without adnexectomy, showed an increased risk of total mortality ( HRs 1.12 95 % CI 1:03 to 1:21 ), lethal and non- lethal cardiovascular disease ( HRs 1.17 95 % CI 1:02 to 1:35 ) and stroke ( HRs 1.14 95 % CI 0.98-1.33 ) (9) . In this population of women subjected to salpingectomy, the surgery wasn't able to lead to an improvement in general survival (10).

Considering the new histopathological classification of the epithelial ovarian cancer, proposed by Kurman (11) and based on new acquisitions about the pathogenesis and the origin of these tumors, it is possible to conceive a new preventive strategy associated with a less morbidity.

In fact, the carcinogenesis model proposed by Kurman, provides for the classification of the most important histological types of epithelial tumors into two types, diversified according to clinico-pathological and genetic features.

The type I is composed of low-grade serous, low-grade endometrioid, clear cell and mucinous carcinomas, whose the ovarian borderline tumors and endometriosis represent the pre-neoplastic lesions. Conversely, the II type includes high-grade endometrioid carcinomas, carcinosarcomas and undifferentiated carcinomas and, more frequently, high-grade serous carcinomas, whose preneoplastic lesion, now, seems to be represented by the serous tubal intraepithelial carcinoma (STIC).

Plenty of evidence, to support the correlation between the epithelial ovarian cancer and the STIC, has been obtained by immunohistochemical and molecular genetics investigations (11). However, from a clinical point of view, this association has been demonstrated only by a study on 55 patients affected by a high-grade serous carcinoma, whose results have shown an involvement in the endosalpinx in 70% of cases and the presence of STIC in about 50% of cases (12).

Some studies, performed on BRCA1 / 2 populations, showed the presence of strongly sites reactive to p53, defined "p53 signature", in the distal tube (13). These sites seem to be more frequent and characteristically multifocal in those tubes with concomitant STIC (14). The finding of "p53 signature" may, therefore, identify an early clonal expansion of the neoplastic proliferation.

This new theory has given the opportunity to prevent this devastating type of cancer by the addition of the prophylactic bilateral salpingectomy (PBS, with the only removal of the tube and the preservation of the ovaries) in all surgical procedures performed in those women with benign diseases once they have accomplished their reproductive desire. The PBS, in place of the current standard procedure (bilateral salpingo-oophorectomy) could reduce the risk of cancer, improving at the same time the quality of life and reducing the risk of premature death due to cardiovascular disease, seen in women subjected to salpingo-oophorectomy before the onset of natural menopause.

Our preliminary data (17) show that, if the bilateral salpingectomy is performed with great care, no patient has negative effects in terms of ovarian function. In addition, in our experience, no perioperative complication is attributable to salpingectomy alone. Despite the retrospective design of our first study, according to the post hoc analysis, these data have shown a significant statistical reliability.

However, the most recent acquisitions assume that also the tissue surrounding the tube seems to give rise to neoplastic sites, so it is conceivable that a greater oncological radicality can be obtained removing the tube and the adjacent structures (mesosalpinx). Now it remains to prove if also the radical technique of prophylactic salpingectomy causes no functional damage to the ovary.

ELIGIBILITY:
Inclusion Criteria:

* Patients subjected to a laparoscopic surgery for a benign gynecologic disease or who require tubal surgical sterilization, once they have accomplished their reproductive desire, and after the acquisition of a written consent for prophylactic salpingectomy and the ovarian preservation.
* Age between 35 and 50 years
* Regular menstruation with intervals between 22 and 35 days

Exclusion Criteria:

* Patients with a family history of ovarian cancer and with a known mutation of the BRCA1/2 genes
* Patients with a current or a past history of cancer
* Patients who don't consent to the prophylactic salpingectomy
* Patients subjected to hysterectomy
* Previous adnexal surgery
* PCOS
* Estrogen-progestin therapy in the 2 months prior to the enrollment
* Acute or chronic pelvic inflammatory disorders
* Malignant gynecological neoplasms
* Prior chemotherapy or radiotherapy
* Autoimmune diseases, chronic, metabolic, endocrine and systemic disorders, including hyperandrogenism, hyperprolactinemia, diabetes mellitus and thyroid disease
* Hypogonadotropic hypogonadism
* Taking medications that can cause menstrual irregularities
* Other clinical conditions

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Ovarian reserve change | One, and 3 months after surgery
  The basal levels of AMH, FSH and estradiol, the antral follicle count (AFC), the ovarian volume, the Vascularization Index (VI), the flow index (FI) and the 'vascular flow index (VFI) in all healthy women over a period of time between the first and fourth day of their menstrual cycle will be assessed.

SECONDARY OUTCOMES:
Operative times | The same day of surgery
Intraoperative blood loss | two hours after the end of surgery
postoperative hospital stay | The day of patient discharge, everage 4 day after surgery
return to the normal activities | two month after surgery
complication rate | The day of patient discharge, everage 4 day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Chair of Obstetrics and Gynecology - University division - UMG, Catanzaro, CZ, Italy

REFERENCES:
- [Background] Morelli M, Venturella R, Mocciaro R, Di Cello A, Rania E, Lico D, D'Alessandro P, Zullo F. Prophylactic salpingectomy in premenopausal low-risk women for ovarian cancer: primum non nocere. Gynecol Oncol. 2013 Jun;129(3):448-51. doi: 10.1016/j.ygyno.2013.03.023. Epub 2013 Apr 2. PMID 23558052
- [Derived] Venturella R, Morelli M, Lico D, Di Cello A, Rocca M, Sacchinelli A, Mocciaro R, D'Alessandro P, Maiorana A, Gizzo S, Zullo F. Wide excision of soft tissues adjacent to the ovary and fallopian tube does not impair the ovarian reserve in women undergoing prophylactic bilateral salpingectomy: results from a randomized, controlled trial. Fertil Steril. 2015 Nov;104(5):1332-9. doi: 10.1016/j.fertnstert.2015.08.004. Epub 2015 Aug 31. PMID 26335129